CLINICAL TRIAL: NCT05105594
Title: Investigation of Causes of Kinesiophobia, Fatigue and Quality of Life in Patients With Lower Extremity Lymphedema
Brief Title: Causes of Kinesiophobia in Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Cansu Sahbaz Pirincci, Phd, Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CSP1
Record Dates: First submitted 2021-10-26; First posted 2021-11-03 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Lymphedema
Keywords: lymphedema, Kinesiophobia
MeSH Terms: conditions — Lymphedema; Kinesiophobia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Active Comparator): People who have lymphedema
  Interventions: Other: survey application
- control group (Active Comparator): healty people
  Interventions: Other: survey application

INTERVENTIONS:
Other: survey application — Fear of movement will be evaluated with the Kinesiophopia Causes Scale. It is a 20-question survey in which the causes of fear of movement are investigated. Functional Evaluation of Treatment of Fatigue Chronic Disease will be assessed by the Fatigue Questionnaire. It consists of 13 questions assessing the level of fatigue during daily activities in the last 7 days. Quality of Life will be assessed by the Lymphedema Quality of Life Questionnaire.
  Other Names: Lymphedema Group

SUMMARY:
In this study, the reason for the fear of movement in patients with lymphedema will be investigated and recommendations will be given to the patients to eliminate it.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-65
* To be diagnosed with lymphedema in the unilateral lower extremity
* Volunteering to work
* Not having orthopedic disorders in the lower extremities

Exclusion Criteria:

* Not volunteering to participate in the research
* Having bilateral lower extremity lymphedema
* Having an active infection
* Having a mental cognitive disorder
* Being unable to communicate and cooperate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Kinesiophopia Causes Scale | 10 minutes
  It is a 20 question survey. A higher score on the questionnaire indicates that they have more fear of movement.
functional assessment of chronic illness therapy | 10 minutes
  It consists of 13 questions assessing the level of fatigue during daily activities in the last 7 days.
Lymphedema Quality of Life Questionnaire | 10 minutes
  It is a survey consisting of 21 questions. High scores indicate lower quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No